CLINICAL TRIAL: NCT01699360
Title: The Biomarker for CYP3A-mediated Immunosuppressive Agents Metabolism in Chinese Renal Transplant Recipients
Brief Title: The Biomarker for Immunosuppressive Agents Metabolism in Chinese Renal Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Xi Luo, clinical research assistant, Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H3110-81072700
Record Dates: First submitted 2012-09-26; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Immunosuppressive Agents; Hydrocortisone; Cortisone
MeSH Terms: interventions — Cyclosporine; Tacrolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclosporine A, Tacrolimus, Sirolimus (Experimental): Cyclosporine A：soft capsule,2-6mg/kg/d, the same twice daily dose at least five days.
  Tacrolimus:capsule,0.15-0.3mg/kg/d, the same twice daily dose at least five days.
  Sirolimus:tablet,2mg/d, once a day.
  Interventions: Drug: Cyclosporine A, Tacrolimus, Sirolimus

INTERVENTIONS:
Drug: Cyclosporine A, Tacrolimus, Sirolimus

SUMMARY:
The aim of this study is to evaluate the potential of endogenous cortisol and cortisone metabolism as a biomarker for immunosuppressive agents disposition in Chinese renal transplant recipients. If the blood concentrations of immunosuppressants can be predicted successfully, this new probe may take place of current drug monitoring post transplantation.

DETAILED DESCRIPTION:
Immunosuppressive agents, including cyclosporine A, tacrolimus, and sirolimus, have been widely used to improve the outcome of organ transplantation. The need for frequent and specific monitoring of drug concentrations remains essential, since the therapeutic dosing and pharmacokinetics show great variability among recipients. However, this may be time and cost consuming. Indeed, cyclosporine A, tacrolimus, and sirolimus are all metabolized by CYP3A, consisting with the metabolic characteristic of endogenous cortisol and cortisone. Hence, the present study is designed to determine if the endogenous cortisol and cortisone metabolism can be used as an noninvasive probe for immunosuppressants pharmacokinetics in Chinese renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adult patients who had undergone their first renal transplantation； All patients received an immunosuppressive regimen containing immunosuppressive agents, mycophenolate mofetil, and corticosteroids; All patients had normal liver and renal function.

Exclusion Criteria:

* an acute rejection episode or infection; multiple organ transplantation; taking any other medications known to interact with immunosuppressive agents, with exception of calcium-channel blockers; abnormal findings on physical examination or laboratory tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The relationship between the ratio of 6β-hydroxycortisol and 6β-hydroxycortisone to cortisol and cortisone in urine and pharmacokinetic parameters of immunosuppressive agents | 0-144h post-dose
  For renal transplant recipients, blood samples are collected at 0 time point (before dosing) for the analysis of trough concentrations of immunosuppressive agents, and urine samples are gathered at 2h interval post-dose (8:00am-10:00am).
  For healthy subjects, blood samples are collected at 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24h after cyclosporine A dosing; at 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72h after tacrolimus dosing; at 0, 0.33, 0.67, 1, 2, 3, 4, 5, 8, 10, 12, 16, 24, 48, 72, 96, 120h after sirolimus dosing. Urine samples are obtained for 0-10 h (8:00 am to 18:00 pm) and 10-24 h (18:00 pm to 8:00 am) post-dose. Furthermore，blood samples at 1, 4, 8, 10, 24h and urine samples for additional 24 h interval (-8:00 am to 8:00 am) before dosing are compared with those obtained after dosing to evaluate the effects of immunosuppressive agents administration on cortisol and cortisone levels and metabolism.

SECONDARY OUTCOMES:
The relationship between plasma 6β-hydroxylation clearance of the sum of cortisol and cortisone and pharmacokinetic parameters of immunosuppressive agents | 0-144h post-dose
  The same as in the Primary Outcome Measure

CONTACTS AND LOCATIONS:
Overall Officials: Zeneng cheng, doctor, Study Director — Central South University
Locations (1):
- The third xiangya hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Cai N, Li B, Huang X, Xu K, Feng H, Cheng Z, Zhu L, Zheng L, Luo X. A non-invasive CYP3A4 biomarker and body mass index predict cyclosporine dosage requirements in Chinese renal transplant recipients. Pharmazie. 2015 Dec;70(12):815-8. PMID 26817280